CLINICAL TRIAL: NCT02731391
Title: Clinical Research on Bowel Symptoms of Patients With Pelvic Organ Prolapse
Brief Title: Clinical Research on Bowel Symptoms of Patient With Pelvic Organ Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Tan Cheng, doctor, Peking University People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pkuph-0103969
Record Dates: First submitted 2016-01-28; First posted 2016-04-07 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Bowel Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesh repairment (Experimental): patients undergoing pelvic floor Reconstruction using mesh
  Interventions: Procedure: Pelvic floor reconstruction（with or without mesh）
- Tradition Neoplasty (Active Comparator): patients undergoing traditional surgical approaches
  Interventions: Procedure: Pelvic floor reconstruction（with or without mesh）

INTERVENTIONS:
Procedure: Pelvic floor reconstruction（with or without mesh）

SUMMARY:
To study the prevalence of bowel symptoms in patients with pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

* The patients with stage>2 POP are recruited.The patients are all received surgeries, which include transvaginal synthetic mesh surgery, the sacral fixation, tissue repair surgery and colpocleisis.

Exclusion Criteria:

* Gestation；
* Inflammatory bowel disease；
* Slow transit constipation diagnosed by Colonic transit test；
* Unable to follow up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
change in the prevalence of bowel symptoms | baseline,1,3,6,12 months after operation.
change in the severity of intestinal symptoms | baseline,1,3,6,12 months after operation.
  assessed by Birmingham Bowel and Urinary Symptoms Questionnaire

SECONDARY OUTCOMES:
change in the quality of life | baseline,1,3,6,12 months after operation.
  assessed by international consultation on incontinence questionnaire short form
length of the high-pressure zone recorded by anorectal manometry | baseline and 12 months after operation
rectoanal inhibitory reflex recorded by anorectal manometry | baseline and 12 months after operation
Rectal-Vaginal pressure interval during maximum Vasalva | baseline and 6 months after operation
  Measured by Peritron manometer

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China